CLINICAL TRIAL: NCT03485352
Title: Influence of the Sleep and Chronotype Pattern in Metabolic, Anthropometric and Biochemical Responses in Patients Submitted to Bariatric Surgery
Brief Title: Influence of the Sleep Pattern in Patients Submitted to Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Cibele Aparecida Crispim, Principal Investigator, Federal University of Uberlandia
Other Study IDs: CEP UFU 2459483/2017
Record Dates: First submitted 2018-02-20; First posted 2018-04-02 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-09

CONDITIONS: Bariatric Surgery Candidate
Keywords: Bariatric Surgery; Sleep; Chronotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bariatric Surgery patients: Patients attending a private clinic specialized in the treatment of obesity and bariatric surgery. Patients to be analyzed should have a medical indication for bariatric surgery.

SUMMARY:
The present study has a prospective, longitudinal and observational character, will be performed with patients attending a private clinic specialized in the treatment of obesity and bariatric surgery. Patients to be analyzed should have a medical indication for bariatric surgery.

DETAILED DESCRIPTION:
The patients will be selected for ten months and will be monitored for 12 months there are preoperative period, 3 months, 6 months and 12 months after surgery. Anthropometrical evaluation, biochemistry, polysomnography and sleep questionnaire (Epworth and Psqi) and midpoint sleep questionnaires will be performed to classify the chronotype for sleep pattern evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study and sign the Informed Consent Form (EHIC)
* Patients submitted to By-pass or Sleeve bariatric surgery or Endossleve
* Patients with BMI above 35 kg / m².
* Over the age of 18 and up to 60 years.

Exclusion Criteria:

* Failure to provide the information necessary for the development of the study.
* Patients undergo revisional surgery

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Bariatric Surgery patients
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cibele A Crispim, PhD, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Cibele Aparecida Crispim, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carvalho AC, Mota MC, Marot LP, Mattar LA, de Sousa JAG, Araujo ACT, da Costa Assis CT, Crispim CA. Circadian Misalignment Is Negatively Associated with the Anthropometric, Metabolic and Food Intake Outcomes of Bariatric Patients 6 Months After Surgery. Obes Surg. 2021 Jan;31(1):159-169. doi: 10.1007/s11695-020-04873-x. Epub 2020 Jul 29. PMID 32728839

RESULTS

PARTICIPANT FLOW:
Groups:
- Bariatric Surgery Patients: Patients undergoing bariatric surgery (sleeve or Bypass) 28 male and 94 woman with mean age of 33 years old.
Period: Overall Study
Arm/Group | Bariatric Surgery Patients
Started | 122 (Baseline)
3 Months | 117 (3 months)
Completed | 113 (6 months)
Not Completed | 9
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Population: Bariatric patients in six months follow - up after surgery
Groups:
- Small SJL: Patients who underwent bariatric surgery - Roux-en-Y gastric bypass (80%) or Sleeve (20%), female (80%)
- Large SJL: Patients who underwent bariatric surgery - Roux-en-Y gastric bypass (79%) or Sleeve (21%), female (74%)
- Total: Total of all reporting groups
Arm/Group | Small SJL | Large SJL | Total
Number analyzed (Participants) | 60 | 62 | 122
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: The participants were categorised as follows: initially, the mean exposure to SJL of the three assessment periods was calculated. Subsequently, the median of this distribution was determined and used to categorise the participants into two groups: large exposure to SJL (mean exposure > median) or small exposure to SJL (mean exposure ≤ median
  years | 33.5 [28 to 39] | 33 [28 to 39] | 33 [28 to 41.7]
Sex: Female, Male [Count of Participants; unit: Participants] — Brazilian bariatric patients
  Participants
    Female | 48 | 46 | 94
    Male | 12 | 16 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Social jetlag exposure [Median (Inter-Quartile Range); unit: Minutes] — The participants were categorised as follows: initially, the mean exposure to SJL of the three assessment periods was calculated. Subsequently, the median of this distribution was determined and used to categorise the participants into two groups: large exposure to SJL (mean exposure > median) or small exposure to SJL (mean exposure ≤ median).
  Minutes | 67 [43 to 107] | 67 [43 to 107] | 67 [43 to 107]

OUTCOME MEASURES:

1. Primary Outcome: Weight in Kg
Description: Anthropometric assessment will be evaluated using weight (kg).
Time Frame: Baseline, 3 and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of weight in the preoperative evaluation and in the third and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: Kg
Groups:
- Small SJL: Patients who underwent bariatric surgery - Roux-en-Y gastric bypass (80%) or Sleeve (20%), female (80%) and aged 33 years old.
- Large SJL: Patients who underwent bariatric surgery - Roux-en-Y gastric bypass (79%) or Sleeve (21%), female (74%) and aged 33 years old.
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
Kg
  Baseline | 111.4 (2.1) | 116.4 (3.3)
  3 months | 89.7 (1.7) | 93.5 (2.7)
  6 months | 77.5 (1.5) | 84.2 (2.6)

2. Primary Outcome: BMI in Kg/m²
Description: Anthropometric assessment will be evaluated using BMI (kg/m²).
Time Frame: Baseline, 3 and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of BMI in the preoperative evaluation and in the third and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: Kg/m²
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
Kg/m²
  Baseline | 40.8 (0.4) | 41.8 (0.8)
  3 months | 32.9 (0.4) | 33.6 (0.7)
  6 months | 28.7 (0.4) | 30.2 (0.7)

3. Primary Outcome: Waist Circumference in Centimeters (cm)
Description: Anthropometric assessment will be evaluated using waist circumference (cm)
Time Frame: Baseline, 3 and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of waist circumference in the preoperative evaluation and in the third and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: Centimeters
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
Centimeters
  Baseline | 109.3 (1.4) | 110.0 (1.7)
  3 months | 94.1 (1.2) | 95.1 (1.4)
  6 months | 85.5 (1.1) | 88.4 (1.4)

4. Primary Outcome: Hip Circumference in Centimeters (cm)
Description: Anthropometric assessment will be evaluated using hip circumference (cm)
Time Frame: Baseline, 3 and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of hip circumference in the preoperative evaluation and in the third and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: Centimeters
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
Centimeters
  Baseline | 128.9 (1.1) | 131.4 (1.7)
  3 months | 114.9 (1.1) | 117.8 (1.7)
  6 months | 105.8 (1.0) | 109.9 (1.6)

5. Primary Outcome: Neck Circumference in Centimeters (cm)
Description: Anthropometric assessment will be evaluated using neck circumference (cm)
Time Frame: Baseline, 3 and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of neck circumference in the preoperative evaluation and in the third and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: Centimeters
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
Centimeters
  Baseline | 39.2 (0.4) | 39.4 (0.5)
  3 months | 36.0 (0.4) | 36.3 (0.4)
  6 months | 34.4 (0.3) | 35.1 (0.4)

6. Primary Outcome: Metabolic Parameters - Fasting Glucose (mg/dl)
Description: Metabolic parameters will be evaluated using fasting glucose (mg/dl)
Time Frame: Baseline and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of fasting glucose in the preoperative evaluation and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
mg/dl
  Baseline | 99.0 (1.7) | 101.2 (3.6)
  6 months | 84.5 (1.1) | 83.3 (0.8)

7. Primary Outcome: Metabolic Parameters - Insulin (mg/dl)
Description: Metabolic parameters will be evaluated using insulin (mg/dl)
Time Frame: Baseline and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of insulin in the preoperative evaluation and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
mg/dl
  Baseline | 27.0 (2.1) | 25.2 (1.6)
  6 months | 8.8 (0.9) | 10.5 (0.6)

8. Primary Outcome: Metabolic Parameters - Homeostasis Model Assessment for Beta-cell Function (HOMA - IR)
Description: Values of metabolic parameters will be evaluated using Homeostasis model assessment for beta-cell function (HOMA - IR) according to the standard assessment measurement in mg/dl. Higher values reflect worse insulin resistance
Time Frame: Baseline and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of HOMA IR in the preoperative evaluation and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
mg/dl
  Baseline | 6.7 (0.5) | 6.2 (0.4)
  6 months | 1.8 (0.2) | 2.1 (0.1)

9. Primary Outcome: Metabolic Parameters - Cholesterol (mg/dl)
Description: Metabolic parameters will be evaluated using Cholesterol (mg/dl)
Time Frame: Baseline and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of cholesterol in the preoperative evaluation and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
mg/dl
  Baseline | 201.6 (5.3) | 203.9 (5.4)
  6 months | 157.0 (4.2) | 159.5 (4.6)

10. Primary Outcome: Metabolic Parameters - High Density Lipoprotein Cholesterol (HDL - mg/dl)
Description: Metabolic parameters will be evaluated using High density lipoprotein cholesterol (HDL - mg/dl)
Time Frame: Baseline and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of HDL in the preoperative evaluation and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
mg/dl
  Baseline | 51.4 (1.7) | 47.6 (1.6)
  6 months | 52.1 (1.6) | 47.1 (1.5)

11. Primary Outcome: Metabolic Parameters - Low Density Lipoprotein Cholesterol (LDL - mg/dl)
Description: Metabolic parameters will be evaluated using low density lipoprotein cholesterol (LDL -mg/dl)
Time Frame: Baseline and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of LDL in the preoperative evaluation and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
mg/dl
  Baseline | 118.0 (4.4) | 119.8 (4.3)
  6 months | 86.0 (3.5) | 92.9 (3.8)

12. Primary Outcome: Metabolic Parameters - Very Low Density Lipoprotein Cholesterol (VLDL - mg/dl)
Description: Metabolic parameters will be evaluated using Very low density lipoprotein cholesterol (VLDL - mg/dl)
Time Frame: Baseline and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of VLDL in the preoperative evaluation and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
mg/dl
  Baseline | 32.2 (2.6) | 36.4 (2.9)
  6 months | 19.3 (0.9) | 19.4 (1.1)

13. Primary Outcome: Metabolic Parameters - Triglycerides (mg/dl)
Description: Metabolic parameters will be evaluated using Triglycerides (mg/dl)
Time Frame: Baseline and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of triglycerides in the preoperative evaluation and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
mg/dl
  Baseline | 162.9 (10.6) | 162.3 (9.0)
  6 months | 98.8 (5.7) | 96.0 (4.6)

14. Secondary Outcome: Food Consumption - Calories (Grams/Day)
Description: The food consumption was evaluated by two 24-h recalls at each evaluation moment (Baseline, third and sixth month), with one occurring on a weekday (applied in a private room with the interviewer and participant only) and the other one on the weekend (applied by phone, as done in previous studies).
Time Frame: Baseline, 3 and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of food consumption of calories in the preoperative evaluation and in the third and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: grams/day
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
grams/day
  Baseline | 2185.0 (95.5) | 2565.6 (130.0)
  3 months | 823.8 (32.0) | 889.7 (34.2)
  6 months | 937.7 (30.6) | 1091.9 (39.0)

15. Secondary Outcome: Food Consumption - Carbohydrate (Grams/Day)
Description: as for outcome 14
Time Frame: Baseline, 3 and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of food consumption of the carbohydrate in the preoperative evaluation and in the third and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: grams/day
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
grams/day
  Baseline | 229.0 (9.4) | 261.4 (13.7)
  3 months | 61 (3.1) | 70.7 (3.7)
  6 months | 68.8 (3.5) | 77.7 (3.8)

16. Secondary Outcome: Food Consumption - Total Fat (Grams/Day)
Description: as for outcome 14
Time Frame: Baseline, 3 and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of food consumption of total fat in the preoperative evaluation and in the third and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: grams/day
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
grams/day
  Baseline | 97.3 (5.6) | 116.5 (7.4)
  3 months | 32.2 (1.7) | 33.2 (1.9)
  6 months | 40.2 (1.7) | 49.5 (2.4)

17. Secondary Outcome: Food Consumption - Polyunsaturated Fat (Grams/Day)
Description: as for outcome 14
Time Frame: Baseline, 3 and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of food consumption of Polyunsaturated fat in the preoperative evaluation and in the third and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: grams/day
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
grams/day
  Baseline | 12.9 (0.9) | 15.9 (1.2)
  3 months | 4.5 (0.2) | 5.0 (0.3)
  6 months | 5.9 (0.3) | 7.8 (0.5)

18. Secondary Outcome: Food Consumption - Monounsaturated Fat (Grams/Day)
Description: as for outcome 14
Time Frame: Baseline, 3 and 6 months
Population: Generalised estimating equations with gamma distribution and adjusted for possible confounding factors were used to examine the effect of SJL exposure level (large or small) between these factors on the evolution of food consumption of Monounsaturated fat in the preoperative evaluation and in the third and sixth months after the surgical intervention.
Measure: Mean (Standard Error); unit: grams/day
Arm/Group | Small SJL | Large SJL
Number analyzed (Participants) | 60 | 62
grams/day
  Baseline | 30.1 (1.9) | 34.5 (1.9)
  3 months | 10.0 (0.6) | 10.2 (0.6)
  6 months | 12.8 (0.5) | 15.6 (0.9)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year and 5 months
Description: The risks are that during blood collection it may eventually be painful for the volunteer causing bruises or swelling caused by blood collection, embarrassment '' shame'' for weight measurement and circumferences and during the application of questionnaires. Adverse events were evaluated and monitored throughout data collection,however none of these situations was identified during the study.
Groups:
- Small and Large Social Jetlag: Patients who underwent bariatric surgery (Roux-en-Y gastric bypass or Sleeve - 77% female, aged 33 years (range 28-41)).
Arm/Group | Small and Large Social Jetlag
All-Cause Mortality (participants affected / at risk) | 0/122
Serious Adverse Events (participants affected / at risk) | 0/122
Other Adverse Events (participants affected / at risk) | 0/122

LIMITATIONS AND CAVEATS:
Use of questionnaires, which, although valid and widely used in others research, are subjective and dependent on the participants' memory.

The participants underwent only two different surgical techniques in a private service.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-04-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03485352/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03485352/SAP_001.pdf
  • Informed Consent Form (2021-04-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03485352/ICF_002.pdf